CLINICAL TRIAL: NCT00483080
Title: NGR006: A Phase II Study of NGR-hTNF Administered as Single Agent Every 3 Weeks or Weekly in Patients Affected by Colorectal Cancer (CRC), Previously Treated With Fluoropyrimidine, Oxaliplatin and Irinotecan Based Regimens
Brief Title: Study of NGR-hTNF as Single Agent in Patients Affected by Colorectal Cancer (CRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR006; 2006-005451-15 (EudraCT Number)
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer (CRC)
Keywords: NGR-hTNF; CRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A: NGR-hTNF (Experimental): NGR-hTNF: 0.8 mcg/m² as 60-minutes intravenous infusion every 3 weeks or weekly
  Interventions: Drug: NGR-hTNF

INTERVENTIONS:
Drug: NGR-hTNF — iv q3W or q1W NGR-hTNF 0.8 μg/m²

SUMMARY:
The main objective of the trial is to document the progression free survival (PFS) in advanced or metastatic colorectal cancer patients treated with NGR-hTNF as single agent. Safety will be established by clinical and laboratory assessment according to NCI-CTC criteria.

DETAILED DESCRIPTION:
This is a phase II, open-label, non-randomized study that will be conducted in patients affected by advanced or metastatic colorectal cancer (CRC), previously treated with fluoropyrimidine, oxaliplatin and irinotecan based regimens, that will be conducted using Simon's two-stage design method.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years affected by advanced or metastatic colorectal cancer (CRC), previously treated with fluoropyrimidine, oxaliplatin and irinotecan based regimens, but not more than three lines of therapy. Adjuvant chemotherapy following definitive management of the primary lesion in the colon or rectum is allowed and will not be counted as a line of therapy

  * ECOG Performance status 0 - 1
  * Patients in progression disease at study entry, CT documented
  * Adequate baseline bone marrow, hepatic and renal function, defined as follows:
* Neutrophils > 1.5 x 10^9/L and platelets > 100 x 10^9/L
* Bilirubin < 1.5 x ULN
* AST and/or ALT < 2.5 x ULN in absence of liver metastases
* AST and/or ALT < 5 x ULN in presence of liver metastases
* Serum creatinine < 1.5 x ULN

  * Absence of any conditions in which hypervolemia and its consequences (e.g. increased stroke volume, elevated blood pressure) or hemodilution could represent a risk for the patient (reference appendix "Technical data sheet human albumin")
  * Normal cardiac function and absence of uncontrolled hypertension
  * Patients must give written informed consent to participate in the study

Exclusion Criteria:

* More than three lines of chemotherapy (except biological agents)
* Concurrent anticancer therapy
* Patients may not receive any other investigational agents while on study
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e.menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | during the study
  PFS evaluated according to Response evaluation criteria in solid tumors (RECIST)

SECONDARY OUTCOMES:
Tumor Growth Control Rate (TGCR) | during the study
  TGCR evaluated according to Response evaluation criteria in solid tumors (RECIST)
Overall survival (OS) | during the study
  Defined as the time from the date of randomization until the date of death due to any cause or the last date the patient was known to be alive
Circulating tumor cells (CTCs) | before and following the treatment
  To document modification of CTCs
Experimental imaging study (DCE-MRI) | before and following the first cycle
  to document possible modifications on vessels permeability
to evaluate AUC(tau) of NGR-hTNF in patients treated with weekly schedule | during the first 6 weeks (time points: prior to infusion, 20 minutes, 60 minutes, 90 minutes, 120 minutes and 240 minutes after treatment start)
  to evaluate AUC(tau) of NGR-hTNF administered weekly
to evaluate Cmax of NGR-hTNF in patients treated with weekly schedule | during the first 6 weeks (time points: prior to infusion, 20 minutes, 60 minutes, 90 minutes, 120 minutes and 240 minutes after treatment start)
  to evaluate Cmax of NGR-hTNF administered weekly
Safety according to NCI-CTCAE criteria (version 3) | during and following the treatment
  To evaluate safety profile related to NGR-hTNF

CONTACTS AND LOCATIONS:
Overall Officials: Federico Caligaris Cappio, MD, Principal Investigator — Fondazione San Raffaele del Monte Tabor
Locations (3):
- Italy (3):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliera Universitaria "San Martino", Genoa
  - Fondazione San Raffaele del Monte Tabor, Milan

REFERENCES:
- [Result] Santoro A, Rimassa L, Sobrero AF, Citterio G, Sclafani F, Carnaghi C, Pessino A, Caprioni F, Andretta V, Tronconi MC, Finocchiaro G, Rossoni G, Zanoni A, Miggiano C, Rizzardi GP, Traversari C, Caligaris-Cappio F, Lambiase A, Bordignon C. Phase II study of NGR-hTNF, a selective vascular targeting agent, in patients with metastatic colorectal cancer after failure of standard therapy. Eur J Cancer. 2010 Oct;46(15):2746-52. doi: 10.1016/j.ejca.2010.07.012. Epub 2010 Aug 12. PMID 20708923